CLINICAL TRIAL: NCT03093779
Title: Mechanisms of Health Literacy and Information Accessibility in the Deaf
Acronym: HIL
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Rochester Institute of Technology (Other); Sinai Health System (Other); Hurley Medical Center (Other); Boston University (Other)
Responsible Party: Principal Investigator, Michael McKee, Assistant Professor of Family Medicine, University of Michigan
Other Study IDs: HUM00104423
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Hearing Loss; Health Literacy
Keywords: Hearing Loss; Deaf; Health Literacy; Health Information; Visual Learning
MeSH Terms: conditions — Hearing Loss; Spatial Learning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deaf: Individuals who are deaf and use sign language to communicate.
  Interventions: Other: Health Information Assessment
- Hearing: Individuals with no hearing loss and who communicate in spoken English.
  Interventions: Other: Health Information Assessment

INTERVENTIONS:
Other: Health Information Assessment — Assess how hearing loss and health literacy alters the ability to access and comprehend online health information

SUMMARY:
The purpose of this proposal is to examine the attitudes, knowledge, and skills related to health information that influence health literacy among Deaf individuals.The study team will also examine frequently overlooked potential predictors of health literacy, including cognitive abilities, resilience, and self-efficacy. To achieve the study objectives, researchers will conduct an explanatory sequential mixed methods design using extensive quantitative data collection procedures, namely, cross-sectional surveys and measures that will identify predictors and moderators of health literacy with Deaf and hearing subjects. These results will inform the subsequent qualitative assessment using elicitation interviews that will help explain the quantitative results, and elucidate how and why Deaf individuals access and understand health information. A community advisory board consisting of Deaf community members will provide oversight to the proposal that will be led by multiple Deaf investigators, including the PI. The Deaf community, due to communication barriers, relative social marginalization, and their reliance on visual learning, provides a unique insight into how health information is distributed and disseminated visually. Findings may be applicable to other individuals with hearing loss who navigate and cope with life more visually than the typical hearing person. This will be critical to determine more accurately the effect of visual learning and existing online health information on health literacy.

DETAILED DESCRIPTION:
University of Michigan(UM) is the clinical coordinating center (CCC) and data coordinating center (DCC) for this study. There are no subject recruitment or interaction will take place at UM. CCC engages clinicians and the clinical research mission and provides the training and professional development to ensure effective study by recruiting and maintaining the study sites performed at the Hurley Medical Center at Flint, Michigan, The National Technical Institute of Technology(NTID) at Rochester Institute of Technology in Rochester, New York, and The Sinai Deaf Health(SDH)program in Chicago, Illinois including participates. Thus, educating and training investigators, study coordinators, and other research staff to ensure an ongoing quality improvement of research processes. DCC is highly invested in producing the highest quality survey questionnaires for use with deaf ASL-users and hearing, English speakers. The study team will only use the best possible ASL translations of the data collection measures in order to best obtain accurate, high-quality research.

University of Michigan (UM) will function as the lead site, not as a performance site. UM will oversee all three other sites and conduct quality checks with each site, assist with training of the staff for standardization, and conduct data management/storage of de-identified data along with analysis. Hard copies and identifiers will be maintained at each site as per their approved IRB protocols.

The two primary objectives of this proposal are:

* To elucidate the role of information marginalization on health literacy in Deaf American Sign Language (ASL) users
* To better understand the mechanisms of health literacy in this population so as to identify viable targets for future health literacy intervention development. This proposal is responsive to PAR-10-133's request for studies that assess mechanisms underlying health literacy, including roles of cognition, culture, language fluency, and information-seeking and interpretation ability in the deaf population and, how these may differ from the hearing population.

A secondary objective is to assess how varying levels of hearing loss can affect individuals' abilities to access and comprehend health information and their health literacy adequacy.

ELIGIBILITY:
Inclusion Criteria:

Deaf American Sign Language Users:

- deaf persons who use sign language and live in Flint, Michigan, Rochester NY, and Chicago, IL metropolitan areas.

Hearing, English speakers:

- hearing persons who speak fluent English and live in Flint, Michigan, Rochester NY, and Chicago, IL metropolitan areas.

Exclusion Criteria:

* Those who have cognitive impairment (e.g., due to dementia, delirium or intoxication).
* Those who unable to consent to the study.
* Individuals with limited vision will be excluded if they are unable to effectively use a PC (i.e., function vision at 20-200 or worse).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 450 Deaf ASL users and 450 Hearing native English speakers
Sampling Method: Non-Probability Sample
Enrollment: 901 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Health Literacy | 5 minutes in a single data assessment
  Use of the American Sign Language- Newest Vital Sign and the English version of the Newest Vital Sign will be used to assess health literacy. Scores range from 0-6 with 5-6 considered to be adequate health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McKee, MD, MPH, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - Mount Sinai Hospital, Chicago, Illinois
  - Hurley Medical Center, Flint, Michigan
  - Rochester Institute of Technology/National Technical Institute for the Deaf, Rochester, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McKee MM, Hauser PC, Champlin S, Paasche-Orlow M, Wyse K, Cuculick J, Buis LR, Plegue M, Sen A, Fetters MD. Deaf Adults' Health Literacy and Access to Health Information: Protocol for a Multicenter Mixed Methods Study. JMIR Res Protoc. 2019 Oct 9;8(10):e14889. doi: 10.2196/14889. PMID 31599730
- [Background] Champlin S, Cuculick J, Hauser PC, Wyse K, McKee MM. Using Gaze Tracking as a Research Tool in the Deaf Health Literacy and Access to Health Information Project: Protocol for a Multisite Mixed Methods Study and Preliminary Results. JMIR Res Protoc. 2021 Sep 7;10(9):e26708. doi: 10.2196/26708. PMID 34491211
- [Result] Panko TL, Contreras J, Postl D, Mussallem A, Champlin S, Paasche-Orlow MK, Hill J, Plegue MA, Hauser PC, McKee M. The Deaf Community's Experiences Navigating COVID-19 Pandemic Information. Health Lit Res Pract. 2021 Apr;5(2):e162-e170. doi: 10.3928/24748307-20210503-01. Epub 2021 Jun 22. PMID 34213997